CLINICAL TRIAL: NCT04340453
Title: The Comparison of Hip and Knee Focused Exercises Versus Hip and Knee Focused Exercises With the Use of Blood Flow Restriction Training in Adults With Patellofemoral Pain: A Randomized Controlled Trial.
Brief Title: The Comparison of Hip and Knee Focused Exercises Versus Hip and Knee Focused Exercises With the Use of Blood Flow Restriction Training in Adults With Patellofemoral Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: European University Cyprus (Other)
Responsible Party: Principal Investigator, Antonis Constantinou, PT, MSc, PhD(can), Department of health Sciences , Physiotherapy Programme, European University Cyprus, Cyprus member of Cyprus Musculoskeletal and Sports Trauma Research Centre (CYMUSTREC), European University Cyprus
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ΕΕΒΚ/ΕΠ/2019/86
Record Dates: First submitted 2020-04-06; First posted 2020-04-09 (Actual); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Patellofemoral Pain Syndrome
Keywords: Patellofemoral Pain; Exercise; Rehabilitation; Blood Flow Restriction training; physical therapy; physiotherapy
MeSH Terms: conditions — Patellofemoral Pain Syndrome; Motor Activity | interventions — Exercise; Blood Flow Restriction Therapy; Papaverine

STUDY DESIGN:
Intervention Model Description: This a randomized controlled trial with first primary end point at four weeks and second primary end point at two months. Participants will be allocated randomly into one of two intervention groups. Group1 (Knee and hip focused exercises) Group 2 (knee and hip focused exercises with BFR)
Who Masked: Investigator, Outcomes Assessor
Masking Description: participants and care providers were only blinded to the other groups intervention.
  The Investigator and outcomes assessor are blinded to patient allocation and data code.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Hip and Knee Exercise Program) (Active Comparator): Standard exercise physiotherapy treatment of a Hip and Knee Exercise Program plus stretching.
  Interventions: Other: Hip and Knee Exercise Program; Other: stretching
- Group 2 (BFR-training hip and knee exercise group) (Experimental): BFR-training hip and knee exercise group plus stretching.
  Interventions: Other: Exercise with Blood Flow restriction training; Other: stretching

INTERVENTIONS:
Other: Exercise with Blood Flow restriction training — 3 times a week for 4 weeks to a total of 12 sessions. BFR cuff (Sports Rehab Tourniquet©) will be used, with a width of 10cm and a length of 116cm or 84cm depending on the diameter of the participants thigh. Therapy sessions will be supervised and in groups. Exercises focus on strengthening the hip extensors and abductors, as well as the quadriceps both in open and closed kinetic chain. Exercises will be carried out using will be set at a load of 30% of 1RM with a limb occlusion pressure (LOP) of 70%. The first set will consist of 30reps. followed by 3 sets of 15reps. at 2:2 (con/ecc) at 60bpm by Metronome app. with auditory cue. Rest between sets will be 30sec and between exercises 2min. Cuffs will be deflated during the resting period between exercises and re-inflated at the beginning of the next exercise. Exercise progression will be individualized based on assessments at the beginning of each week. The duration has been estimated to be approximately 60min. including LOP estimation.
  Other Names: BFR training
  Arms: Group 2 (BFR-training hip and knee exercise group)
Other: Hip and Knee Exercise Program — A supervised hip and knee strengthening exercise protocol with a combination of stretching, 3 times a week for 4 weeks to a total of 12 sessions. Exercises focus on hip extensors, abductors, as well as the quadriceps and hamstrings strength. Open Kinetic Chain (OKC) exercises will be executed first followed by CKC exercises. Exercises using weights or mechanical resistance will be set at a load of 70% of 1RM and 3 sets of 10 rep. for each exercise. Elastic band exercises will be set at 10RM for 3 sets. Tempo will be set by the Metronome app installed on a Smartphone at 1:2 (con/ecc) at 60bpm with auditory cue. Rest between sets will be 30sec and between exercises 2min. Exercise progression will be individualized based on assessments at the beginning of each week. The duration of each session is estimated to be approximately 45min, with the exception of the first session of each week which is estimated to be 80min due to the addition of strength testing
  Other Names: Standard treatment
  Arms: Group 1 (Hip and Knee Exercise Program)
Other: stretching — Both groups will receive stretching of the hamstrings, plantar flexors, quadriceps and Iliotibial Band (ITB) in the same manor at the end of each session. Passive stretching will be executed by the physiotherapist with 3x30sec stretch for each muscle group

SUMMARY:
Hip and Knee strengthening exercises are implemented in Patellofemoral Pain (PFP) rehabilitation but exercising in high loads to achieve muscle changes in strength may lead to increased patellofemoral joint stress. Low load training with Blood Flow Restriction (BFR) may allow for exercise strength benefits to proximal and distal muscles with reduced joint stress and by promoting hypoalgesia.

The purpose of this study is to compare hip and knee focused exercises with and without BFR training in adults with PFP. The main outcome of this study is function ability which will be measured with the Kujala Anterior Knee pain Scale translated in the Greek language at four weeks post intervention and at two months follow up. Our null hypothesis is that there will be no difference between groups for primary and secondary outcomes measured at four weeks and two months post intervention.

DETAILED DESCRIPTION:
This a randomized controlled clinical trial with first primary end point at four weeks and second primary end point at two months.

Sample size was determined through power analysis. The Minimal Clinically Significant Difference (MCID) of our main outcome measure, Kujala Anterior Knee Pain Scale, was used for the estimation. The MCID of the Kujala scale has been reported to be 10 points with an estimated standard deviation of 13,5 points. For a power of 0.80 and a level of significance a=0.05 and considering a two tailed t-test the sample size was calculated to be 60 participants total (30 in each group). The GPower 3.0.10 software was used to calculate the sample size. By estimating a possible 20% drop out we concluded to a sample size of 75.

The participants of this study will be volunteers and considered a sample of convenience since no official records or data base exists in Cyprus with all PFP patients. Participant recruitment will begin in November 2019. Potential participants will be informed for the study through printed posters around the European University Cyprus (EUC) campus, local social media online posters and will volunteer for inclusion. Screening will be carried out by an orthopedic surgeon, at the musculoskeletal laboratory of the EUC to determine their eligibility based on specific inclusion and exclusion criteria.

Volunteers who meet inclusion criteria will receive oral and written information and give informed consent to participate in the study by signing a consent form. They will be randomized into one of two treatment groups. Group 1 will be the Hip and Knee Exercise group and Group 2 the BFR training Hip and Κnee exercise group. Randomization will be carried out using a block sequence of 4 by an external statistician to maintain a balance in sample size across groups over time and to ensure the assessor was blind to the participants allocation.

All interventions will take place in the musculoskeletal laboratory and the training center lab of the EUC. Time consistency in treatments will be a goal, in order to train participants at similar circadian rhythm. Room temperature for both labs will be set at 25 °C. Two experienced physiotherapists will each be randomly assigned to supervise one of the two intervention groups and provide the treatment. The therapists role is to supervise treatments and their progression, keep track of compliance with the study design, adverse effects and drop outs. If patients do not comply with the study (seek other treatment for PFP, exercise during the study, inability to attend treatments) design they will be excluded. The two therapist will be blinded as to the other groups treatment protocol and the studies outcomes. They will be given written information for all procedures of their intervention group in order to ensure consistency throughout the study. Data collected by the therapists will be stored at the E.U.C laboratories and will only be available to them. Additionally, the therapists will be assisted by fourth year physiotherapy undergraduate students in supervising participants during treatments. Participants who fail to complete at least 10/12 therapy sessions will be excluded and their data will not be analyzed. All therapy sessions will be supervise by a physician who will be in charge of participants safety. Any adverse events will be reported with publication of final results. Participants are free to withdraw from the study at any given moment. In case of any complaints, participants have the right to file official complaints to the university bioethics committee.

Planed statistical analysis: Statistical analysis will be performed by the studies assessor who is blinded to the participants treatment group using the IBM SPSS "Statistical Package for the Social Sciences" (SPSS, Version 20.0). Descriptive statistics will be analyzed with the calculation of means, standard deviations, minimum and max values for each variable. A normality check will follow using the One Sample Kolmogorov-Smirnov test (p<0.05). The chi-squared test will be used to test for difference between the two groups with respect to the categorical variable gender. To check for differences within groups (baseline-4weeks, baseline-2months follow up and 4weeks-2months follow up) we will use the paired t-test for each comparison. In case of nonparametric data, the Wilcoxon signed rank test will be used. In order to estimate differences between the two groups (baseline-4weeks, baseline-2months follow up and 4weeks-2months follow up) we will use the mixed two way ANOVA with time as a within-subjects factor and treatment as the between subjects factor. Homogeneity of variance will be checked with the Levene test <0.05. In the case of not normally distributed data we will use the generalized mixed effect model with treatment as a fixed factor, time as a random factor, and inverse as the link function. Possible correlations will also be checked for our outcome measures using the Pearson correlation coefficient. In case of not normally distributed data the Spearman correlation coefficient will be used if there seems to be a linear correlation from a scatter plot. Missing values in the Patient Reported Outcome Measures will be imputed using Multiple Imputation (MI). Only upon agreement by the authors that there will be no further changes and/or analysis, results of the study will be published.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers to be included can be either male or female, must be 18-40 years of age and should have at least a 4 week, history of peri or retro-patella non traumatic pain, with intensity of worst pain during the previous week at 3cm on the Visual Analogue Scale (VAS).
* Pain should be aggravated by at least two of the following functional tasks: squatting, kneeling, prolonged sitting, stair ascending or descending, hopping or running.
* During physical examination pain must be present with either palpation of the patella facets or with the patella compression test or a deep squat.
* Volunteers with bilateral symptoms will be documented but the limb with the worst pain will be used for analysis.

Inclusion criteria are based on latest PFP guidelines

Exclusion Criteria:

* Athletes will be excluded, as well as participants with a high level of physical activity based on assessment of the International Physical Activity Questionnaire (IPAQ) in Greek. This will be performed on the day of initial screening. Their exclusion is based on the fact that they may not respond to the level of intensity of the exercises provided in this study and for homogeneity of the sample.

Volunteers with the following characteristics will also be excluded:

* History or current meniscus ligament or other knee injury and/or surgery.
* Other knee pathology such as knee osteoarthritis, Osgood- Schlatter or Sinding-Larsen-Johanssen syndrome or tendinopathy of muscles surrounding the knee. Knee instability, feeling of "giving way", history of subluxation or dislocation of the knee joint or joint edema.
* Extended use of NSAID or cortisone.
* Referred pain from lumbar spine or another region.
* Patella dysplasia, rheumatoid arthritis or neurological syndromes or diseases
* During clinical examination volunteers with pain located on the patella tendon that is eliminated with isometric contraction, the pes anserinus, the Iliotibial Band (ITB), or with a positive medial or lateral patella apprehension test will also be excluded
* Volunteers that had previous treatment for PFP in the past 6 months will also be excluded to avoid non responders and carryover effects from previous treatments.
* Volunteers with unexplained chest pains
* Cardiovascular disease, renal disease, vascular surgery or disease
* Deep Venous Thrombosis (DVT) or high risk for DVT, resent surgery ≤6 months, - High blood pressure (≥140/90mmHg) dizzy spells, history of fainting or dizziness with exercise
* Pregnancy
* Any contraindication to exercise

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2019-11-29 (Actual); Primary Completion 2019-12-21 (Actual); Study Completion 2020-02-29 (Actual)

PRIMARY OUTCOMES:
"change" is being assessed for Function The Greek version of the Kujala Anterior Knee Pain Scale (AKPS) | baseline, 4 weeks (end of treatment), 2 months (follow up)
  The AKPS is a 13-item questionnaire that documents response to six different activities such as walking, running, jumping, stair climbing, squatting and prolonged sitting with knee bent, as well as patients symptoms, such as limping, inability to weight bear on the affected limb, swelling, abnormal patella movement, muscle atrophy and limitations of flexion of knee joint. The AKPS asks about the duration of symptoms and limb(s) affected. The maximum score is 100 (no pain/disability/limitation) and the minimum 0 (worst possible function). This questionnaire has been previously used in PFP studies and is found to be a valid and reliable measure for PFP patients with a minimally clinical significant difference (MCID) of 10points. The Greek version has been found to have good internal consistency (Cronbach's a=0.942), test-retest reliability (ICC=0.921) and concurrent validity (r>0.7)

SECONDARY OUTCOMES:
"change" is being assessed. Pain with the Visual Analog Scale | baseline, 4 weeks (end of treatment), 2 months (follow up)
  Pain will be assessed using the visual analog scale VAS 0-10cm. This scale is a 10cm horizontal line with two small vertical lines at the two ends. The far-left side is 0 "no pain" and the far right is 10 "worst pain". Participants will be asked to mark with a horizontal line to rate the level of worst pain VAS-W and the level of their usual pain VAS-U that they experienced during the course of the previous week. A standard ruler will be used to measure the distance from 0 to the participants mark. The VAS scale measuring these two types of pain have been shown to be valid and reliable in patients with PFP with an MCID of 2cm.
"change" is being assessed. Pain with single leg squatting (shallow-deep) | baseline, 4 weeks (end of treatment), 2 months (follow up)
  Two depths of squatting will be assessed and the VAS scale will be used to quantify the level of pain with each squat. For the first Single-leg squat (shallow): the participant will stand in front of the treatment bed and the height of the bed will be adjusted to be the mid-point of his thigh (halfway between the greater trochanter and popliteal fossa midpoint). For the second Single-leg squat (deep): the beds height will be adjusted to the popliteal fossa midpoint. Participants will perform the squat with hands crossed over the chest until they touch but not sit on the beds surface. At the end of each test, the VAS scale will be used to measure pain felt during the squat. This testing method has been previously used to assess pain in anterior knee pain patients.
"change" is being assessed. Kinesiophobia: The Tampa scale of Kinesiophobia (TSK) | baseline, 4 weeks (end of treatment), 2 months (follow up)
  We will assess Kinesiophobia using the Greek Version of the TSK that has been found to be valid and reliable. This scale consists of 17 items that assess fear of injury due to movement. Participants will be asked to make ratings of their degree of agreement for each of the 17 items. Ratings range from 1 (strongly disagree) to 4 (strongly agree). Responses will be summed after reversing the scores of items 4,8,12 and 16. Higher total scores relate to higher related fear.
"change" is being assessed. Catastrophizing: The Pain Catastrophizing Scale (PCS) | baseline, 4 weeks (end of treatment), 2 months (follow up)
  The Pain Catastrophizing Scale (PCS) assesses the cognitive process by which pain is seen as an extreme threat and from which the patient suffers exaggerated negative consequences. We will assess catastrophizing using the Greek Version of the PCS that has been found to be valid and reliable. The questionnaire consists of 13 items (statements) describing pain experience and participants are asked to indicate whether they agree with these statements on a five point scale rating from 0 (not at all) to 4 (always). Scores are summed to calculate a final score. A high score indicates a high level of pain catastrophizing. The PSC measures three categories: rumination, magnification and helplessness. Rumination refers to the patients' inability to apart the pain from his mind, magnification expresses the exaggerated cognitions of pain as a threat, and hopelessness is the estimation that the patient cannot do anything to influence his pain.
"change" is being assessed. Maximum pain free flexion angle using the decline step down test | baseline, 4 weeks (end of treatment), 2 months (follow up)
  This is a functional test that measures the Maximum Pain Free Flexion Angle (MPFFA) of the knee joint whilst descending a 20cm high step with a surface inclination of 20o. The participant descends from the step to the maximum point where no pain is present. At this point the assessor will take a photo using the Dr. Goniometer (DrG) app, installed on an iPhone 6S andmeasure the MPFFA. The test has been found to be reliable with intra-observer reliability ICC=0.83 and inter-observer reliability ICC=0.85. It has been shown to be valid as it has been correlated with the AKPS (r= 0.31, p= 0.030
"change" is being assessed. Strength: Strength tests will measure isometric Maximum Voluntary Contraction (MVIC) with the use of a MicroFET2TM Hand Held Dynamometer (HHD). | baseline, 4 weeks (end of treatment), 2 months (follow up)
  Strength tests will measure isometric Maximum Voluntary Contraction (MVIC) with the use of a MicroFET2TM Hand Held Dynamometer (HHD) for the quadriceps at ≈60o of knee flexion from the seated position. Hip extensors will be assessed from the prone position and hip abductors in the side-lying position with the hip abducted to ≈10o. Strength will be recorded in Newtons (N). Testing will begin after 2-3 sub-maximal contractions for familiarization and warm up followed by a maximal isometric contraction of a 5sec duration with standard verbal encouragement by the assessor. then followed by a 30sec rest and then repeated. If the two measures differ less than 10% then no other testing will follow. The mean of the two measures will be used for analysis. If measures differ >10%, a third test will be repeated until the above criteria is met. Placement of the dynamometer will be marked with a marker to ensure consistency between trials.

CONTACTS AND LOCATIONS:
Overall Officials: Antonis Constantinou, PhDcan, Principal Investigator — European University Cyprus; Dimitris Stasinopoulos, PhD, Study Director — European University Cyprus
Locations (1):
- European University Cyprus, Nicosia, Engomi, Cyprus

IPD SHARING:
Plan to Share IPD: Yes
Only upon agreement by the authors that there will be no further changes and/or analysis, results of the study will be published and shared. No patient data will be shared to be compliant with the latest GDPR code.
Supporting Information: Study Protocol, CSR
Time Frame: 6 months after publication date and only upon agreement by the authors that there will be no further changes and/or analysis may data be shared.
Access Criteria: It is to the authors discretion to share study data to other researchers.